CLINICAL TRIAL: NCT07096440
Title: NOVo-Helisen Depot HoUSe Dust Mites - A Prospective, Multicenter, Noninterventional Clinical Study on the Tolerability and Safety of Short One Strength UP-dosing in Children, Adolescents, and Adults in Daily Practice
Brief Title: Noninterventional Study on Tolerability and Safety of One Strength Updosing With Novo-Helisen Depot House Dust Mites
Acronym: NOVUS-UP
Status: Not yet recruiting | Type: Observational
Sponsor: Allergopharma GmbH & Co. KG (Industry)
Responsible Party: Sponsor
Other Study IDs: AL2501NH
Record Dates: First submitted 2025-07-17; First posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Allergic Rhinitis Due to House Dust Mite; Allergic Conjunctivitis Due to Dermatophagoides Farinae; Allergic Conjunctivitis Due to Dermatophagoides Pteronyssinus; Allergic Asthma Due to Dermatophagoides Farinae; Allergic Asthma Due to Dermatophagoides Pteronyssinus
Keywords: Allergen Immunotherapy; Allergopharma; Novo-Helisen Depot; Allergy; House Dust Mites; One Strength; NHD (D.p./D.f.); NHD; Children; poland; SCIT
MeSH Terms: conditions — Hypersensitivity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this non-interventional study is to investigate the safety and tolerability of a new simplified up-dosing schedule for Novo-Helisen Depot.

Novo-Helisen Depot is an approved allergen immunotherapy used to treat allergies to house dust mites. For allergen immunotherapy, it is important that the allergen dose is gradually increased, a process known as up-dosing to induce immune tolerance to the allergen. The recently approved One Strength up-dosing scheme for Novo-Helisen Depot allows up-dosing with 6 injections instead of the previously required 14 injections.

The main questions the study aims to answer are:

How is the tolerability and the safety of One Strength up-dosing scheme in daily practice? This study includes approximately 105 patients (children (≥5 years), adolescents, and adults), receiving this treatment as part of their usual care.

Study data on safety and tolerability wil be collected for each patient during the first 8 injection visits.

The study will be conducted at 6-8 study sites in Poland.

DETAILED DESCRIPTION:
The Standard dose escalation scheme with the unmodified (native) SCIT house dust mite preparation Novo-Helisen Depot consists of 14 injections.

The newly approved One Strength dose escalation scheme, recently approved for children (≥5 years), adolescents (12-17 years) and adults (≥18 years), offers a simplified dose escalation scheme with only 6 injections. To date, the safety and tolerability of this One Strength escalation scheme has been demonstrated in 2 clinical trials involving 243 patients (aged 5-65 years). The objective of the present non-interventional study is to compare the safety and tolerability of the One Strength dose escalation scheme (6 injections) in different age groups (children, adolescents, adults) and to supplement available clinical trial data on safety and tolerability with clinical study data in daily practice.

Data collection during the first 8 visits of treatment with NHD (D.p./D.f.) using the One Strength dose escalation scheme:

Visit 1: Informed consent, In-/Exclusion-criteria, demographics, medical history, first injection (dose escalation)

Visits 2-6: 2nd to 6th injection (dose escalation)

Visits 7-8: 7th and 8th injection (maintenance doses)

In line with the SmPC recommendations, all patients must be monitored for at least 30 minutes after each injection and then be examined by the physician. Individually, this observation time may be prolonged.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent from the patient. For patients under the age of 18, the consent of both parents/legal guardians is also required.
* Patients who are eligible for treatment with the One Strength dose escalation scheme of NHD (D.p./D.f.) according to the specifications in the SmPC. These include children (5 to <12 years), adolescents (≥12 to <18 years) and adults (≥18 years) with allergic (IgE-mediated) diseases, such as allergic rhinitis, allergic conjunctivitis, allergic bronchial asthma (see section 4 of the current SmPC)
* The treatment decision must precede the decision to participate in the study and must be independent.

Exclusion Criteria:

* Any contraindication according to section 4.3 of the current SmPC for NHD (D.p./D.f.) for the One Strength dose escalation scheme.

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This NIS will enroll a total of 105 patients, including 35 children (aged ≥5 to < 12 years), 35 adolescents (aged ≥12 to <18 years), and 35 adults (aged ≥ 18 years).
  Patient recruitment will be conducted at six to eight allergy-specialized study sites across Poland.
  Participation in this NIS follows the independent and prior decision by the treating physician and the patient to begin therapy with the One Strength dose escalation scheme of NHD (D.p./D.f.). The indication and use of the One Strength up-dosing scheme of NHD (D.p./D.f.) is based exclusively on the individual therapeutic need.
Sampling Method: Non-Probability Sample
Enrollment: 105 (Estimated)
Dates: Start 2025-07-30 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Safety of the One Strength dose escalation scheme in daily practice | up to study completion, approximately 11 to 20 weeks
  * Number, incidence, type, intensity and time of occurrence of (serious) adverse events ((S)AEs)
  * Number, incidence, type, intensity and time of occurrence of (serious) adverse drug reactions ((S)ADRs)
  * Frequency and intensity of systemic allergic reactions
  * Proportion of patients who reach the maintenance dose without/with dose adjustment
Tolerability of the One Strength dose escalation scheme in daily practice | up to study completion, approximately 11 to 20 weeks
  Tolerability will be assessed by both the treating physicians and the patients using a 5-point Likert scale (Likert, 1932) with the following categories: "Very bad," "Bad," "Average," "Good," and "Very good".

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Dr. med. Marek Jutel, Principal Investigator — "ALL-MED" Specjalistyczna Opieka Medyczna. Medyczny Instytut Badawczy

IPD SHARING:
Plan to Share IPD: No